CLINICAL TRIAL: NCT05591495
Title: The Role of Laparoscopy in Upper Abdominal Surgical Emergencies in Adults: A Retrospective Observational Study.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: zagazig university 12
Record Dates: First submitted 2022-10-07; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Acute Abdomen
Keywords: Emergency surgery; Laparoscopy; Upper abdominal surgery
MeSH Terms: conditions — Abdomen, Acute | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopy in upper abdominal surgical emergencies in adults — evaluation the role of laparoscopy in upper GIT emergencies in adults

SUMMARY:
Introduction Laparoscopy can be used to diagnose and treat the etiologies of acute abdominal pain. This study aimed to assess laparoscopy's effectiveness in upper gastrointestinal (G.I.T) emergencies regarding intra-and postoperative outcomes.

Method: A retrospective observational study was conducted in the emergency departments of Zagazig University on 215 patients who had upper abdominal emergency surgeries between June 2017 and June 2020.

DETAILED DESCRIPTION:
When surgical procedures are standardized, laparoscopy's benefits in a range of emergency scenarios are without question acknowledged. When only a basic strategy is set for the surgery, and the surgical approach entirely depends on intra-abdominal findings, the benefits are diminished or unknown. The evidence unequivocally supports the superiority of a laparoscopic approach in numerous emergency cases, such as acute cholecystitis, gastroduodenal perforated ulcers, infected pancreatic necrosis, and splenic injuries Laparoscopy gives the primary advantages of a shorter hospital stay, a quicker procedure, and faster recovery without complications. Rapid recovery is connected with early enteral feeding. Adequate nutritional support aids in maintaining homeostasis and, as a result, enhances immunity, thereby decreasing the incidence of wound infection. Laparoscopy should be considered with caution whenever abdominal access is considered difficult, as in cases of organ enlargement, adhesion, and bowel distension. In actuality, creating the pneumoperitoneum is an essential step in the procedure. Increased intraperitoneal pressure produces cardio-respiratory and neurological effects.

In this study, the investigators designed a retrospective observational study to present our experience in assessing the outcomes of a laparoscopic approach in emergent upper abdominal surgery in terms of intraoperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnoses of upper G.I.T. emergencies, namely acute cholecystitis, perforated P.U., acute necrotizing pancreatitis, and splenic trauma.

Exclusion Criteria:

* < 18 years of age and
* open surgeries for upper G.I.T.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Between June 2017 and June 2020, 215 patients were admitted to Zagazig University Hospital's emergency surgical unit with clinical diagnoses of upper G.I.T. emergencies, namely acute cholecystitis, perforated P.U., acute necrotizing pancreatitis, and splenic trauma. The work has been reported following STROBE guidelines. To be included in the study, patients must meet the following criteria: >18 years of both sexes complaining of acute upper G.I.T. emergencies and undergoing laparoscopic surgeries, namely acute cholecystitis, perforated peptic ulcer, pancreatic necrosis, and splenic injuries. < 18 years of age and open surgeries for upper G.I.T. emergency surgeries were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
intraoperative complications requiring conversion | 2 years
  the number of patients converted to open approach

SECONDARY OUTCOMES:
postoperative complications requiring reintervention | within 2 years of surgery
  reintervention

IPD SHARING:
Plan to Share IPD: No